CLINICAL TRIAL: NCT00269932
Title: A Multicenter, Randomized Study to Compare the Safety and Efficacy of Oral Levofloxacin With That of Cefuroxime Axetil in the Treatment of Acute Bacterial Exacerbation of Chronic Bronchitis in Adults
Brief Title: A Study of the Safety and Effectiveness of Oral Levofloxacin Compared With Cefuroxime Axetil in the Treatment of Adults With Persistent Bronchitis Experiencing Rapid Onset of Severe Worsening of Symptoms Caused by Bacteria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005497
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-02

CONDITIONS: Bronchitis, Chronic
Keywords: Bronchitis; chronic bronchitis; lung diseases; respiratory tract infections; bronchial diseases; antibacterial agents; quinolones; levofloxacin
MeSH Terms: conditions — Bronchitis, Chronic; Bronchitis; Lung Diseases; Respiratory Tract Infections; Bronchial Diseases | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of levofloxacin, an antibiotic, compared with cefuroxime axetil, another antibiotic, in the treatment of adults with chronic bronchitis experiencing rapid onset of worsening of symptoms caused by bacteria.

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel group, multicenter study to determine the safety and effectiveness of 500 mg of levofloxacin (once daily for 5 - 7 days) compared with 250 mg of cefuroxime axetil (every 12 hours for 10 days) in adults with chronic bronchitis experiencing rapid onset of severe worsening of symptoms caused by bacteria. The study consists of 3 visits: one visit for screening and enrollment, and 2 visits for assessment of safety and effectiveness (one visit on Days 3 - 5 of the study and one visit [post-therapy] 5 - 7 days after the last dose of the study drug). The total duration of patient participation in the study is approximately 2 weeks. The primary efficacy assessment is the clinical response 5 - 7 days after the last dose of study drug, (categorized as cured, improved, or failed) based upon changes in signs and symptoms. Safety evaluations (incidence of adverse events, physical examination, laboratory tests) are performed throughout the study. The study hypothesis is that treatment with levofloxacin is at least as effective and as well tolerated as treatment with cefuroxime axetil in adult patients with chronic bronchitis experiencing sudden worsening of symptoms caused by bacterial infection. Levofloxacin 500 mg by mouth once daily for 5 - 7 days, or cefuroxime axetil 250 mg by mouth every 12 hours for 10 days

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic obstructive lung disease (chronic bronchitis and/or emphysema) with rapid onset of worsening of symptoms caused by bacterial infection
* recent increase in cough
* change in type or amount of sputum (the mucus produced on coughing)
* findings during the physical examination of clinical signs and symptoms of chronic obstructive lung disease
* received previous antibiotic treatment if the previous treatment lasted for 24 hours or less, or if the previous treatment lasted longer than 24 hours but there was no improvement or stabilization of the disease.

Exclusion Criteria:

* Illness requiring antibiotic treatment by injection into a vein, beneath the skin, or into a muscle, or patient has a requirement for a second antibiotic medication taken orally in addition to the study drug
* infection due to bacteria known (prior to the start of the study) to be resistant to the study drugs
* previous allergic or serious adverse reaction to antibiotics similar to the study drugs
* diagnosis of pneumonia determined by x-ray at the start of the trial
* has cystic fibrosis, seizure disorders, kidney disease, or an unstable psychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 1993-08; Study Completion 1994-05 (Actual)

PRIMARY OUTCOMES:
Clinical response rate (reduction in signs and symptoms) at post-therapy (5 - 7 days after the last dose of study drug)

SECONDARY OUTCOMES:
Rate of elimination of disease-causing bacteria, by patient, and by type of bacteria; incidence of adverse events; changes in physical examination and laboratory tests after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the safety and effectiveness of levofloxacin taken by mouth compared with cefuroxime axetil in the treatment of adults with persistent bronchitis experiencing rapid onset of severe worsening of symptoms caused by bacteria — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=658&filename=CR005497_CSR.pdf